CLINICAL TRIAL: NCT04573634
Title: A Registry Study of COVID-19 Serologic and Virologic Testing to Accelerate Recovery and Transition (START) - Assessment of COVID19 Penetrance in HCW and Non HCW in Kentucky
Brief Title: A Registry Study of COVID-19 Serologic and Virologic Testing to Accelerate Recovery and Transition
Acronym: START
Status: Withdrawn | Type: Observational
Why Stopped: Low accrual
Sponsor: Jill M Kolesar (Other)
Responsible Party: Sponsor-Investigator, Jill M Kolesar, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: PHARM-20-COVID19-START
Record Dates: First submitted 2020-09-30; First posted 2020-10-05 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Covid19; SARS-CoV Infection
Keywords: prevalance; risk-factor; population; Kentucky; antibody; SARS CoV-2; seroconversion; physical distancing; PCR; quarantine
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal swabs, whole blood, serum, plasma and buffy coat
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Health Care Workers: Health-care workers undergoing standard of care assessment of SARS-CoV-2 serology testing at UKHC.
- Eligible Patients: Patients undergoing standard of care assessment of SARS-CoV-2 serology testing at UKHC.
- Quarantining Individuals: Individuals with a COVID-19 exposure requiring quarantine who are asymptomatic and who will receive standard of care SARS-CoV-2 PCR testing.

SUMMARY:
The co-primary objectives of this study are to:

1. Determine and compare the COVID-19 antibody positivity rate in health care workers and patients without a known COVID-19 infection
2. Determine if PCR negativity for COVID-19 early in quarantine predicts negativity at Day 14 in quarantining individuals

DETAILED DESCRIPTION:
This is a prospective cohort study designed to identify the prevalence of IgG antibodies to SARS CoV-2 as well as to assess risk factors for IgG positivity. It will compare rates of positivity and risk factors among healthcare workers and non-healthcare workers and assess the ability of PCR negativity at day 3 or 4, 5, 7, or 10 to predict negativity on day 14 in individuals quarantining after a COVID exposure.

In addition to having a standard of care clinical antibody test, both healthcare workers, quarantining individuals, and patients will be asked to fill out a survey to assess risk factors for COVID infection and provide a research blood sample. Quarantining individuals will also have standard of care PCR testing on days 3 or 4, 5, 7, 10, and 14 of the quarantine period.

Collected blood samples will be used to assess for the presence of neutralizing antibodies and measure antibodies with a research test. An annual blood specimen and survey will be collected from each study participant for up to 2 years total after study entry.

ELIGIBILITY:
Inclusion Criteria:

* Individuals (health-care workers and patients) undergoing standard of care assessment of SARS-CoV-2 serology testing
* Individuals with a COVID-19 exposure requiring quarantine who are asymptomatic and who will receive standard of care SARS-CoV-2 PCR testing.
* Able to understand and sign the Informed Consent and Research Authorization From.

Exclusion Criteria:

* Prisoners
* Patients with psychiatric illness that would limit compliance
* Patients with social situations that would limit compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals (health-care workers and patients) undergoing standard of care assessment of SARS-CoV-2 serology testing at the University of Kentucky or individuals with a COVID-19 exposure requiring quarantine who are asymptomatic and who will receive standard of care testing. Notably, these individuals may not have active COVID infection; they will be assessed for antibodies which is evidence of a prior, asymptomatic COVID infection or infection associated with a known exposure as diagnosed by polymerase chain reaction (PCR).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of COVID-19 | 2 years
  Proportion of people with IgG antibodies against SARS CoV-2 using a standard of care, Clinical Laboratory Improvement Amendments (CLIA), IgG antibody test.

SECONDARY OUTCOMES:
PCR Conversion in Exposed Individuals | 14 days
  Determine the average time point at which PCR conversion occurs following exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Kolesar, PharmD, MS, Principal Investigator — University of Kentucky; Derek Forster, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No